CLINICAL TRIAL: NCT02861131
Title: The Effect of Sugammadex Versus Neostigmine on Postoperative Pulmonary Complications in Patients 70 Years or Older and Scheduled for 3 Hour or Longer Surgery-A Randomized Controlled Trial
Brief Title: The Effect of Sugammadex Versus Neostigmine on Postoperative Pulmonary Complications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Brandon M Togioka, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MISP #55196
Record Dates: First submitted 2016-07-14; First posted 2016-08-10 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Complications; Neuromuscular Blockade
Keywords: Sugammadex; Neuromuscular Blockade
MeSH Terms: conditions — Postoperative Complications | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Experimental): Sugammadex 2 mg/kg IV once at the end of surgery
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): Neostigmine 0.07 mg/kg to a maximum of 5 mg (+ Glycopyrrolate 0.1-0.2 mg per 1 mg of Neostigmine administered) IV once at the end of surgery
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — At the end of the surgical procedure at a depth of neuromuscular blockade after the reappearance of T2 on the train-of-four, Sugammadex will be dosed once at 2 mg/kg through an intravenous line with brisk flow
  Other Names: Org 25969; Bridion
  Arms: Sugammadex
Drug: Neostigmine — At the end of surgical procedure at a depth of neuromuscular blockade after the reappearance of T2 on the train-of-four, Neostigmine will be dosed once at 0.07 mg/kg to a maximum of 5 mg through an intravenous line with brisk flow. Glycopyrrolate will be administered with Neostigmine at a dose between 0.1 to 0.2 mg of Glycopyrrolate per 1.0 mg of Neostigmine administered.
  Other Names: Prostigmin; Vagostigmin
  Arms: Neostigmine

SUMMARY:
Substantial respiratory morbidity has been associated with postoperative residual paralysis, which is fairly common after general anesthesia involving a neuromuscular blocking agent. Common practice in United States is to reverse neuromuscular blockade with neostigmine at the end of surgery. A new drug with evidence of more complete neuromuscular reversal has been developed, sugammadex. The objective of this study is to determine if a strategy of rocuronium neuromuscular reversal with sugammadex will reduce the proportion of subjects with any postoperative pulmonary complication, compared to neostigmine.

DETAILED DESCRIPTION:
This study is designed to be an assessor-blinded, randomized, controlled, single center, parallel design trial at Oregon Health and Science University (OHSU) in Portland, Oregon. The investigators will enroll patients ≥ 70 years of age that are mentally competent to consent for anesthesia with a scheduled surgical length of ≥ 180 minutes on Monday through Friday in the South Operating Room Theatre at Oregon Health and Science University.

Subjects will be screened for inclusion in the study on either the day prior or the day of surgery. The initial review will occur by a quick view of the surgical posting sheet for the South Operating Rooms. Subjects undergoing any type of surgery will be eligible as long as neuromuscular paralysis is a component of the planned anesthetic. If subjects initially seem appropriate for inclusion, a more in depth chart review will occur. The research coordinator will approach patients that meet inclusion criteria in the Pre-operative Care Unit. Initially all patients 70 years of age or older will have equal probability of being approached for the study. At the halfway point of the study the investigators will monitor enrollment, and if ahead of schedule, preferentially select older patients in the 2nd half of the study-a group that is more likely to have Postoperative Pulmonary Complications (PPCs).

All subjects that are approached for recruitment will hear a description of the study, reasons for pursuing this research question, options for opting out the research protocol or not completing data collection, and potential risks, advantages, and disadvantages from participating. Subjects that agree to participate in the study will be asked to sign a written informed consent that has been approved by our Institutional Review Board. All subjects that agree to participate in the research study will be given a form describing the research study and providing contact information for the principal investigators. The subject's status in the research project will show up clearly on our medical records in their problem list, until the subject's time of participation is complete. A progress note will be placed in the subject's chart to allow other providers to easily contact study investigators. In addition, an electronic copy of the signed consent will be scanned into the medical records system and a copy of the signed consent will be made available for the subject to take home.

All subjects enrolled will have the following characteristics recorded by the research coordinator: age, sex, weight, body mass index, American Society of Anesthesiologists physical status classification score, creatinine clearance, and Charlson comorbidity index.

Subjects will be allocated to either neuromuscular reversal with sugammadex or neostigmine. Before study activation a sample of 200 sequentially numbered opaque envelopes will be prepared by an investigator not involved in patient recruitment, allocation, consent, or assessment: 100 for the sugammadex arm and 100 for the neostigmine arm. Patient allocation will occur in the operating room when the anesthesia provider notifies the coordinator that reversal is appropriate. At that time the research coordinator will open the lowest remaining numbered free envelope. Group assignment will be determined by a computer generated random number sequence produced in Excel (Redmond, Washington). The random number sequence will be generated by an investigator not involved in either patient enrollment or patient assignment. Reversal of rocuronium neuromuscular blockade (i.e. sugammadex or neostigmine) will be defined in the opened opaque envelope. Once a study subject signs a consent form, a unique number corresponding to the opened opaque envelope will be assigned to that subject. The envelope will not be opened until the anesthesia provider is ready to prepare and administer reversal of neuromuscular blockade. This subject number will never be reused and will remain with the subject for the entirety of the study. No subject will ever be allowed to have more than one unique subject number.

The subject, anesthesia providers, and research coordinator performing consent and recruitment will not be blinded to the study drug. The anesthesiologists will not be blinded for reasons of patient safety. The assessor of PPCs, residual neuromuscular blockade, secondary outcomes, exploratory outcomes, and adverse event accounting will be blinded to study drug and will not be allowed in the operating room during surgery.

All subjects will have standard American Society of Anesthesiologists monitors plus five lead electrocardiogram applied. Additional monitoring needs will be left up the anesthesia team directing patient care. Decisions with regards to induction and maintenance of anesthesia will also be left up to the direction of the anesthesia team with the exception that rocuronium will be mandated for maintenance of neuromuscular blockade. Decisions on when to dose and what quantity of rocuronium should be dosed for maintenance of neuromuscular blockade will be left to the discretion of the anesthesia team in the operating room. The level of neuromuscular blockade will be monitored in the operating room at the adductor pollicis muscle with a basic peripheral nerve stimulator monitor that does not have train-of-four ratio capability. Train-of-four counts will be mandated every 15 minutes, which is our current practice at OHSU. Anesthesia providers will be asked to maintain neuromuscular blockade at a T2 level throughout surgery and reverse neuromuscular blockade at as close to a T2 level as safely possible. Administration of sugammadex or neostigmine will occur into a fast flowing IV that is running wide open. Sugammadex will be dosed at 2 mg/kg and neostigmine will be dosed at 0.07 mg/kg to a maximum of 5 mg. Glycopyrrolate will be co-administered in the neostigmine arm at a dose between 0.1 to 0.2 mg of glycopyrrolate per 1.0 mg of neostigmine administered.

In accordance with standard of practice at OHSU, all subjects will have convective warmers used during the case and subject temperature will be monitored. Ventilation parameters will be left to the discretion of the anesthesia team in the operating room.

A train-of-four ratio will be obtained in all subjects within 5 minutes of arrival to the Post-Anesthesia Care Unit (PACU) with a Train-of-four Watch-SX Acceleromyograph. In order to measure the train-of-four ratio in the PACU the train-of-four watch will be set up and calibrated on the subject upon arrival in the OR, prior to the administration of any neuromuscular blocking agent. The accelerometer sensor will be attached to the subject's thumb. The subject's fingers and forearm adjacent to the thumb attached to the accelerometer sensor will be fixed with tape to an arm board to minimize artifact. Ulnar nerve stimulation of the adductor pollicis muscle will be measured via the Train-of-four watch. As twitch height will vary from subject to subject, a control twitch height value of 100% for the 1 Hz mode will be calibrated after a 5 second, 50 Hz tetanic stimulation. This calibration will be used to obtain a train-of-four ratio upon 5 minutes of arrival to the PACU. A train-of-four ratio of less than 0.9 will be considered residual neuromuscular blockade.

Active monitoring of adverse events (desaturation, hypoxemia, upper airway obstruction, aspiration pneumonitis, bronchospasm, laryngospasm, drug hypersensitivity reaction, and recurarization) will be conducted on an ongoing basis until discharge with daily assessments by the research coordinator and/or principal investigator. Assessment of PACU phase 1 recovery time will occur on Post-operative day (POD) #0 or POD #1. Assessment of hospital length of stay will be assessed within a week of discharge by electronic medical record review. Hospital readmission data will be assessed within 1 to 2 months of hospital discharge. National Surgical Quality Improvement Program (NSQIP) 30-day postoperative risk-adjusted respiratory complications will be assessed and recorded prior to data analysis at the conclusion of patient enrollment and study implementation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Elective surgery Monday through Friday in the South Operating Rooms of Oregon Health and Science University (OHSU)
* Planned general endotracheal anesthesia
* Expected surgical duration ≥ 3 hours

Exclusion Criteria:

* Prisoners
* An inability to consent for surgery or anesthesia
* Surgery for which neuromuscular blockade is contraindicated (e.g. neurosurgical, orthopedic, and head and neck surgery in which nerve monitoring will be employed)
* A known neuromuscular disorder
* Stage 4 chronic kidney disease or worse (estimated glomerular filtration rate < 30 ml/min)
* Liver Disease
* An allergies to Sugammadex, Rocuronium, Neostigmine, or Glycopyrrolate
* Patients taking Toremifene

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Togioka BM, Yanez D, Aziz MF, Higgins JR, Tekkali P, Treggiari MM. Randomised controlled trial of sugammadex or neostigmine for reversal of neuromuscular block on the incidence of pulmonary complications in older adults undergoing prolonged surgery. Br J Anaesth. 2020 May;124(5):553-561. doi: 10.1016/j.bja.2020.01.016. Epub 2020 Mar 2. PMID 32139135

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (4.3) | 75.1 (4.0) | 74.9 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 56 | 108
  Male | 48 | 44 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 97 | 93 | 190
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Postoperative Pulmonary Complication
Description: A composite outcome which includes any of the following: postoperative pneumonia, aspiration pneumonitis, atelectasis, pneumothorax, desaturation/hypoxemia, upper airway obstruction, or acute respiratory insufficiency
Time Frame: Length of hospitalization, an average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
Participants | 33 | 40

2. Secondary Outcome: Number of Participants With Residual Neuromuscular Blockade in the PACU
Description: Residual neuromuscular blockade will be defined as a train-of-four ratio < 0.9 taken within 5 minutes of subject arrival in the PACU
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
Participants | 9 | 46

3. Secondary Outcome: PACU Phase 1 Recovery Time
Description: Defined as duration of time required to attain pain control and stable respiratory, haemodynamic, and neurological status
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
minutes | 97.3 (54.3) | 110.0 (62)

4. Other Pre Specified Outcome: Hospital Length of Stay
Description: Defined as the number of days between hospital admission and discharge
Time Frame: Length of hospitalization, an average of 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
days | 4.0 (3.4) | 4.5 (5.0)

5. Other Pre Specified Outcome: Number of Participants With Hospital Readmission Within 30 Days
Description: The proportion of patients that require hospital readmission for any cause within 30 days of hospital discharge
Time Frame: Length of hospitalization plus 30 days post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
Participants | 5 | 15

6. Other Pre Specified Outcome: Number of Participants Diagnosed With a National Surgical Quality Improvement Program (NSQIP) Defined Respiratory Complication
Description: pneumonia, unplanned re-intubation for any reason other than a return trip to the operating room, and ventilator times greater than 48 hours - excluding operating room time
Time Frame: Length of hospitalization, an average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 100 | 100
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 30 days after discharge from the hospital
Arm/Group | Sugammadex | Neostigmine
All-Cause Mortality (participants affected / at risk) | 2/100 | 1/100
Serious Adverse Events (participants affected / at risk) | 2/100 | 3/100
Other Adverse Events (participants affected / at risk) | 50/100 | 52/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=100) | Neostigmine (N=100)
Significant Residual Neuromuscular Paralysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Significant residual Neuromuscular paralysis putting oxygenation and ventilation at risk
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia leading to death (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=100) | Neostigmine (N=100)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 7 (7) | 7 (7)
Nausea or Vomiting (Gastrointestinal disorders) | 14 (14) | 17 (17)
Itching (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8)
Foul, salty or metallic taste (Gastrointestinal disorders) | 19 (19) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02861131/Prot_SAP_000.pdf